CLINICAL TRIAL: NCT07021742
Title: BioHealx® Anal Fistula Device Post Market Surveillance Study
Status: Recruiting | Type: Observational
Sponsor: Signum Surgical USA Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SP002
Record Dates: First submitted 2025-06-02; First posted 2025-06-15 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Fistula-in-ano
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- BioHealx: Subjects will have their anal fistula treated with the BioHealx Anal Fistula Device.
  Interventions: Device: BioHealx

INTERVENTIONS:
Device: BioHealx — Subjects will have their anal fistula treated with the BioHealx Anal Fistula Device, a bioabsorbable implant designed to securely close the fistula internal opening, preventing reinfection, while allowing for drainage through the external opening during healing.

SUMMARY:
This post market surveillance study is a single arm multicenter study to demonstrate the long-term durability and effectiveness of the BioHealx Anal Fistula Device for fistula-in-ano closure (internal and external fistula openings).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years
* Presence of Single Continuous Anal Fistula presenting for initial curative surgery
* Failed or Recurrent Anal Fistula Closure
* Minimum of 6-weeks of draining seton placed prior to procedure.
* Availability for follow-up contacts and willingness to complete the Informed Consent.

Exclusion Criteria:

* Fistula tract shorter than 2cm
* Complex fistula tract (branching)
* Body Mass Index > 35
* Known uncontrolled diabetes or other systemic condition associated with impaired healing
* Known HIV-positive or immunocompromised
* Rectal prolapse
* Pregnancy
* Rectal / fistula malignancy
* Crohn's disease
* Ulcerative proctitis
* Hidradenitis suppurativa of the anal region
* Pilonidal sinus disease
* Presence of hemorrhoid Involving fistula site
* Continuous use of anti-inflammatory
* Intersphincteric fistula in ano or fistula treatable by simple fistulotomy
* Active infection or abscess involving fistula site
* Known allergy to PLGA material
* Any severe acute or uncontrolled chronic disease that according to the investigator might render the patient unsuitable for the study
* Treatment with an investigational drug or medical device in the past 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for treatment of mature, cryptogenic, transsphincteric, non-branching fistulas in ano via tissue apposition.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Successful Closure Repair | 12 Months
  Successful closure repair of the anal fistula as determined by complete healing, i.e., internal and external opening closed (no evidence of an external opening present) without drainage
Non-Recurrence Incidence | 24 and 36 Months
  Non-recurrence incidence determined by continued closure of the external fistula opening.

SECONDARY OUTCOMES:
Fecal Incontinence Quality of Life | 6 Months, 9 Months, 12 Months, 24 Months, 36 Months
  Fecal incontinence Quality of Life (FIQL) score at each follow-up visit (baseline visit and from 6-month and at subsequent follow-up visit) The FIQL score includes 29 items which form four scales: lifestyle, coping/behavior, depression/self-perception, and embarrassment. The FIQL scale range includes a range of response options across its items, from 1 to 4 for most items, 1 to 5 for one item, and 1 to 6 for another. Lower scores indicate lower quality of life.
Fecal Incontinence Severity Index (FISI) | 6 Month, 9 Month, 12 Month, 24 Month, 36 Month
  Fecal Incontinence Severity Index (FISI) at each follow-up visit (baseline visit and from 6-month and at each subsequent follow-up visit).
  The Fecal Incontinence Severity Index (FISI) Scale typically ranges from 0 to a maximum value 61. Higher scores on the FISI scale indicate a worse outcome, reflecting greater severity of fecal incontinence symptoms.
Health Related Quality of Life | 6 Months, 9 Months, 12 Months, 24 Months, 36 Months
  SF-36 Quality of life data will be collected (baseline visit and from 6-month and at each subsequent follow-up visit). Short Form 36 (SF-36) is a generic self-reported outcome measure that quantifies the quality of life in relation to health status. It is a 36-item valid and reliable evaluation with eight areas covering physical functioning, role limitations brought on by physical issues, bodily pain, general health perceptions, vitality, social functioning, role limitations brought on by emotional issues, and perceived mental health. The SF-36 also contains a single question called "health transition" that measures how respondents feel their over health status has changed over the course of a year. The scores range from 0-100 (the worst possible to the most possible)
Pain Score | 6 Months, 9 Months, 12 Months, 24 Months, 36 Months
  Wong-Baker FACES Pain scores will be recorded at each follow-up visit (baseline visit and from 6-month and at each subsequent follow-up visit). The FACES Pain Scale ranges from 0 (no pain) to 10 (the worst pain).
Rescue Analgesic and Therapeutic Antibiotic Use | 6 Weeks, 3 Months, 6 Months, 9 Months, 12 Months, 24 Months, 36 Months
  Occurrence of use of rescue analgesic and/or therapeutic antibiotics beyond post-operative Day 5 after the surgery and at each follow-up visit.

OTHER OUTCOMES:
Device and Procedure Related Adverse Events | 6 Weeks, 3 Months, 6 Months, 9 Months, 12 Months, 24 Months, 36 Months
  Measurement of device and/or procedure related adverse events will be recorded.
Adverse Event Comparison | 6 Weeks, 3 Months, 6 Months, 9 Months, 12 Months, 24 Months, 36 Months
  Measurement of, incidence, severity and persistence of device and/or procedure related adverse events will be recorded and compared with previous BioHealx Anal Fistula Device clinical results and relevant comparator devices (e.g. cutting seton) and procedures (e.g., LIFT).
Occurrence of Fecal Incontinence | Baseline, 6 Weeks, 3 Months, 6 Months, 9 Months, 12 Months, 24 Months, 36 Months
  Fecal continence will be measured through combination of the patient reported Fecal Incontinence Quality of Life questionnaire (FIQL) and the Fecal Incontinence Severity Index questionnaire (FISI) scores at baseline and subsequent periods.
  Fecal incontinence Quality of Life (FIQL) score at each follow-up visit (baseline visit and from 6-month and at subsequent follow-up visit) The FIQL score includes 29 items which form four scales: lifestyle, coping/behavior, depression/self-perception, and embarrassment. The FIQL scale range includes a range of response options across its items, from 1 to 4 for most items, 1 to 5 for one item, and 1 to 6 for another. Lower scores indicate lower quality of life.
  The Fecal Incontinence Severity Index (FISI) Scale typically ranges from 0 to a maximum value 61. Higher scores on the FISI scale indicate a worse outcome, reflecting greater severity of fecal incontinence symptoms.
Rescue Analgesic and Therapeutic Antibiotic Comparison | 6 Weeks, 3 Months, 6 Months, 9 Months, 12 Months, 24 Months, 36 Months
  Rescue analgesic and therapeutic antibiotic use will be recorded and compared with previous BioHealx Anal Fistula Device clinical results and other relevant fistula treatments.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Colorectal Institute, Fort Myers, Florida
  - Maininle Health Lankenau, Bryn Mawr, Pennsylvania

IPD SHARING:
Plan to Share IPD: No